CLINICAL TRIAL: NCT03423901
Title: Impact of Anti-HLA Donor-specific Antibodies in ABO-incompatible Kidney Transplantation
Acronym: A3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/17/0426
Record Dates: First submitted 2018-01-19; First posted 2018-02-06 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Kidney Transplant
Keywords: Complications
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABO/HLA incompatible KT (Experimental): Blood sampling for descriptive analysis of clinical, biological and histological of 12 ABO and HLA incompatible kidney transplantation (KT)
  Interventions: Other: Blood sampling
- ABO incompatible KT (Experimental): Blood sampling for descriptive analysis of clinical, biological and histological of 28 ABO incompatible kidney transplantation
  Interventions: Other: Blood sampling
- HLA incompatible KT (Experimental): Blood sampling for descriptive analysis of clinical, biological and histological of 20 HLA incompatible kidney transplantation
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Descriptive analysis of clinical, biological and histological of 3 arms: ABO incompatible, HLA incompatible, and ABO/HLA incompatible kidney transplantation (1 and 5 years posttransplantation in each groups)

SUMMARY:
It was previously suggested an improvement of graft survival in ABO/HLA incompatible kidney transplantation (KT) compared with HLA (human leukocyte antigen) incompatible transplantation. Here, the investigators would analyse clinical, biological and histological results of ABO/HLA incompatible kidney transplant recipients, comparing with ABO or HLA compatible kidney transplantation.

DETAILED DESCRIPTION:
The investigators propose to analyze the clinical, biological and histological course of kidney function, but also to investigate the T and B cells population after KT in ABO incompatible, ABO/HLA incompatible and HLA incompatible kidney transplantation (1 and 7 years posttransplantation in each groups).

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving a KT and followed at least one year in Toulouse Hospital
* Patient who have signed informed consent
* > 18 years old

Exclusion Criteria:

* Patient under protective measures
* Patients treated for cancer, infectious or immune disease by molecules that could interfere with lymphocyte populations : Interleukin 6 (IL6) blockers, Programmed cell death 1(PD1) and the cytotoxic T-lymphocyte-associated antigen 4 (CTL4) blockers.
* Immunosuppressive treatments withdrawal - Patient in chronic dialysis
* Ongoing pregnancy or pregnancy in the past year
* Past of splenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Gene expression related to antibody mediated rejection | 1 year posttransplantation
  To determine expression of genes related to antibody mediated rejection (inflammation, and endothelial cell activation) by transcriptomic analyse (whole genome micro-array) on kidney biopsies

SECONDARY OUTCOMES:
description of T subsets cells | 1 to 5 years posttransplantation
  to analyse of T subsets cells after Kidney transplantation in blood samples of patients by flow cytometry
description of B subsets cells | 1 to 5 years posttransplantation
  to analyse of B subsets cells after Kidney transplantation in blood samples of patients by flow cytometry
description of lymphocytes rates | 1 to 5 years posttransplantation
  to analyse rates of lymphocytes after Kidney transplantation in blood samples of patients by flow cytometry
Evolution of creatinine clearance | 1 to 5 years posttransplantation
  to analyse creatinine clearance in blood samples of patients after kidney transplantation
Evolution of systematic annual kidney biopsies | 1 to 5 years posttransplantation
  To analyse the evolution of systematic annual kidney biopsies by microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud DEL BELLO, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No